CLINICAL TRIAL: NCT05359120
Title: A Nationwide Multicenter, Ambispective Real-world Study of Pyrotinib Combined With Capecitabine in Patients With HER-2 Positive Advanced Breast Cancer and Brain Metastases (Post-PERMEATE)
Brief Title: Pyrotinib Combined With Capecitabine in HER-2 Positive Advanced Breast Cancer and Brain Metastases (Post-PERMEATE)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HNCH-MBC09-BM03
Record Dates: First submitted 2022-04-29; First posted 2022-05-03 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: HER-2 positive advanced breast cancer; pyrotinib; capecitabine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cohort A: new brain metastases directly treated with pyrotinib combined with capecitabine
- cohort B: whole brain radiotherapy or stereotactic radiotherapy concurrently (≤3 months before and after radiotherapy) with pyrotinib combined with capecitabine
- cohort C: after whole brain radiotherapy or stereotactic radiotherapy (more than 3 months after radiotherapy) treated with pyrotinib combined with capecitabine

SUMMARY:
This study aims to describe the different treatment time, treatment mode and clinical outcomes of pyrotinib maleate tablets combined with capecitabine in the treatment of patients with HER-2 positive advanced breast cancer with brain metastases.

DETAILED DESCRIPTION:
This study is a multicenter, observational, real-world study with no formal statistical assumptions and sample size calculations; patient efficacy and safety data will be descriptively analyzed to assess the risk of HER2-positive advanced breast cancer patients with brain metastases. Efficacy of pyrotinib combined with capecitabine regimen in the real world, while evaluating the overall survival benefit of local therapy and drug therapy in patients with brain metastases.

The estimated sample size is 300 cases, and at least one group of cohort A, cohort B and cohort C is planned to exceed 100 cases; Cohort A - patients with new brain metastases directly treated with pyrotinib combined with capecitabine; Cohort B- Whole brain radiotherapy or stereotactic radiotherapy concurrently (≤3 months before and after radiotherapy) with pyrotinib combined with capecitabine; Cohort C - group of patients with pyrotinib plus capecitabine after whole brain radiotherapy or stereotactic radiotherapy (more than 3 months after radiotherapy)。

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed patients with HER-2 expression-positive advanced breast cancer; Note: Positive HER2 expression refers to at least one tumor cell immunohistochemical staining intensity of 3+ or fluorescence in situ hybridization [FISH] in the pathological detection/recheck of the primary or metastatic lesions performed by the pathology department of the participating central hospital confirmed positive;
2. Brain metastases are diagnosed by MRI/enhanced CT imaging, according to RECIST 1.1 criteria, with or without measurable lesions and with or without symptoms of brain metastases;
3. Pyrotinib combined with capecitabine in the treatment of brain metastases with non-PD evaluation at the first treatment, at least ≥ 2 continuous imaging reports or assessments
4. For previous treatment regimens, no previous use of capecitabine or progression after capecitabine discontinuation for 6 months, or progression after discontinuation of capecitabine adjuvant therapy for one year or more;
5. There are traceable medical history data.

Exclusion Criteria:

1. Patients enrolled in the previous PERMEATE study;
2. The research program is receiving other anti-tumor drug treatment at the same time;
3. The initial dose of pyrotinib is lower than the minimum dose in the instructions (240 mg), and the capecitabine is 50% lower than the standard dose;
4. Pyrotinib combined with capecitabine in the treatment of non-brain metastases and progressive patients;
5. The investigator believes that the patient is not suitable to enter this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases of patients with brain metastases from HER2-positive advanced breast cancer who received pyrotinib combined with capecitabine from July 2018 to December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Time to Failure(TTF) | up to 2 years
  Time from initiation of study protocol treatment to treatment failure or study protocol discontinuation for any reason (including discontinuation due to patient request, disease progression, adverse events, or death)

SECONDARY OUTCOMES:
Progression-free survival(PFS) | up to 2 years
  Time from initiation of study protocol treatment to disease progression (if occurring within 30 days of end of treatment) or death, as assessed by clinician or with or without radiographic progression.
CNS-DCR | up to 2 years
  The patients began to receive the treatment plan of this study, and during the period of the patients' disease progression group, the number of patients with the best response effect of intracranial lesions in the patient's medical records were objective remission (CR+PR) and stable disease (SD) in the analysis data set. The sum of the percentages of the total population.
CNS-CBR | up to 2 years
  The patient started to receive the treatment plan of this study, and during the period of the patient's disease progression group, the best response effect of intracranial lesions in the patient's medical records was complete remission (CR) + partial remission (PR) + stable disease (SD) ≥ 6 The sum of the month's patient population as a percentage of the total population in the analyzed dataset.
CNS-ORR | up to 2 years
  Among all patients who received pyrotinib plus capecitabine for brain metastases, the proportion of patients with physician-assessed complete remission (CR) or any less than complete remission (documented remission) in the patient's medical records on radiology scans.
CNS-DOR | up to 2 years
  Duration between first scan showing documented remission of intracranial lesions and first scan showing disease progression or end of treatment if no progression occurred. rwDOR was evaluable in patients who received ≥2 consecutive radiology scans.
Overall Survival(OS) | up to 2 years
  The time from the start of treatment with this study protocol to the time of all-cause death of patients.
safety | up to 2 years
  Refers to the proportion of patients with a clinically significant adverse event (AE) (ie, leading to treatment modification or discontinuation, patient hospitalization, death, or permanent sequelae) documented in the medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification are available following article publication
Supporting Information: Study Protocol
Time Frame: Three years from publication
Access Criteria: Please contact Central contact person by Email